CLINICAL TRIAL: NCT03951922
Title: Exploring the Effect of Occupational Therapy and Horticulture for Cancer Survivors With Chronic Pain
Brief Title: Occupational Therapy and Horticulture for Cancer Survivors With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Julie Kugel, Program director of Occupational Therapy Doctorate Program, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5180419
Record Dates: First submitted 2019-04-16; First posted 2019-05-16 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Cancer Survivor; Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic Horticulture Group (Experimental): The therapeutic horticulture group will participate in a 6-week horticulture program meeting twice a week for an hour led by an occupational therapist incorporating plant-based activities and education on pain management techniques at a community farm.
  Interventions: Behavioral: Horticultural activity

INTERVENTIONS:
Behavioral: Horticultural activity — Therapeutic horticulture activities are plant-related activities that include but not limited to digging, watering, planting, weeding, trimming, fertilizing, mulching, harvesting, learning about organic farming, and exploring options to incorporate horticulture into daily activities

SUMMARY:
The purpose of this quasi-experimental study is to explore the impact of a therapeutic horticulture program as an occupation-based intervention to address chronic pain symptoms for cancer survivors. The main objectives are to assess participants' perceptions of pain, physical and psychosocial wellness, stress management, and quality of life at pre-, post-, and 3-month follow-up. Quantitative and qualitative data will be synthesized and analyzed to explore this phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 64 years of age
* History of cancer diagnosis
* Chronic pain longer than 3 months
* Have interest in therapeutic horticulture and exercise
* Able to participate in a moderate physical activity in sitting and/or standing for at least one hour twice a week
* Able to provide own transportation to the horticulture site or the supervised exercise program
* Able to comprehend, speak and write in English

Exclusion Criteria:

* Uncontrolled seizure disorder
* Pregnancy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2019-06-08 (Actual); Primary Completion 2019-11-23 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Salivary Cortisol Test | Change between baseline and three months
  Participant stress level will be determined by salivary cortisol levels. Participant's salivary cortisol level will be measured at awakening, 30 minutes following awakening and bedtime. Typically, there is Cortisol Awakening Response (CAR), which is a steep rise in cortisol output during the first 30 minutes following awakening, followed by a steady decline across the morning, afternoon, and evening hours, with the daily nadir typically occurring around midnight. Flattened diurnal cortisol slope relates to increased emotional and psychosocial stress and related to worse health outcomes.
  The typical Cortisol Awakening Response (CAR) is defined as an increase of at least 2.5 nmol/l from the cortisol level taken at awakening. Although there are no agreed norms for the absolute concentrations of free cortisol in saliva it typically ranges between 4.7-18.5 nmol/l for post-awakening, between 8.6-21.9 nmol/l for 30 minutes post-awakening, and 0.3-15.2 nmol/l for bedtime.

SECONDARY OUTCOMES:
Lower body strength | Change between baseline and three months
  Chair Stand testing measures the strength of the lower body. Average scores for this testing are 15 reps for women and 16 reps for men.
Upper body strength | Change between baseline and three months
  Arm Curl testing measures the strength of the upper body. Average scores for this testing are 16 reps for women and 19 reps for men.
Endurance | Change between baseline and three months
  2 Minutes Step testing measures the endurance or physical stamina. Average scores for this testing are 91 times for women and 101 times for men.
Lower body flexibility | Change between baseline and three months
  Chair Sit and Reach testing measures lower body flexibility, specifically your hamstring flexibility. Average scores for this testing are +2 inches for women and + 0.5 inches for men.
Upper body flexibility | Change between baseline and three months
  Back Scratch testing measures the flexibility of the upper body. Average scores for this testing are -0.5 inches for women and -3.5 inches for men.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Kugel, OTD, Principal Investigator — Loma Linda University Health
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No